CLINICAL TRIAL: NCT04317716
Title: A Self-management Program to Prevent Falls in Ambulatory and Non-ambulatory Community Dwelling People With Multiple Sclerosis
Brief Title: A Self-management Program to Prevent Falls in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Charlotte Ytterberg, associate professor (docent), Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-00457
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Feasibility Studies; Accidental Falls; Self-management; Complex Intervention; Group-based; Online Intervention; Short Message Service
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Participants will be stratified for ambulation level (ambulatory/non-ambulatory) and a 1:1 allocation ratio of blocks of 4 will be used.
Who Masked: Outcomes Assessor
Masking Description: The facilitators of the fall prevention program will not be involved in the usual care of the participants. The intervention will take place online. Control-group participants will receive a brochure about falls and fall risk factors, sent by mail. Baseline and follow-up assessments will be performed by blinded evaluators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Fall prevention program and brochure about falls and fall risk factors
  Interventions: Behavioral: fall prevention program
- Control (Other): Bbrochure about falls and fall risk factors
  Interventions: Other: Brochure about falls and fall risk factors

INTERVENTIONS:
Behavioral: fall prevention program — The intervention consists of the fall prevention program for ambulatory and non-ambulatory people with multiple sclerosis. The program will be group-based with 6-8 participants, led by a facilitator, and performed online. It comprises six two-hour sessions held once a week, and a booster session held eight weeks after the sixth session. In addition they will receive a brochure about falls and fall risk factors.
  Arms: Intervention
Other: Brochure about falls and fall risk factors — Control-group participants will receive a brochure about fall risk factors and fall prevention in addition to the standard MS care and rehabilitation.
  Arms: Control

SUMMARY:
This project's overall aim is to develop, deliver, and evaluate feasibility of a fall prevention program for ambulatory and non-ambulatory people with multiple sclerosis. The program will use a comprehensive intervention approach to address a variety of fall risk factors, and utilise self-management strategies. Specific aims are to

1. develop a fall prevention program, that addresses diverse fall risk factors and utilises self-management strategies, for ambulatory and non-ambulatory people with multiple sclerosis using a co-design process.
2. To examine feasibility, acceptability, fidelity, and potential outcome of the online, co-designed self-management fall prevention intervention for ambulatory and non-ambulatory people with multiple sclerosis, and to examine feasibility of the recruitment process, the data collection procedures, and the outcome measures.

DETAILED DESCRIPTION:
Falls among people with multiple sclerosis (PwMS) are common and associated with injuries, fear of falling and low health-related quality of life. Considerations of behavioural, environmental, psychological and physical influences (including ambulation status) are needed to meet fall prevention needs for PwMS. Thus, using a codesign process involving key stakeholders a novel online self-management fall prevention intervention will be created specifically for ambulatory and non-ambulatory PwMS.

The feasibility, acceptability, fidelity and outcome of this complex intervention will be explored. Findings will inform a future full-scale randomised controlled trial. A mixed-method design will be used. Forty-eight PwMS, stratified for ambulation level, will be randomised to control (n=24) or intervention (n=24). Both groups will receive a brochure about fall risk factors and fall prevention. The intervention is group-based (eight PwMS in each group); will be delivered online; and involve six, 2-hour weekly sessions and a booster session 8 weeks after the sixth session. Each intervention group will be led by a trained facilitator.

Data collection will be performed at baseline, and after seven and 18 weeks. Outcome measures will capture data on fall prevention behaviours, fear of falling, falls self-efficacy, social and everyday activities, perceived impact of MS and number of falls. Feasibility of recruitment process, data collection procedures, outcome measures, and delivery, and intervention acceptability, fidelity and outcomes will be evaluated. Both quantitative and qualitative methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged ≥ 18 years
* Diagnosed with multiple sclerosis
* Able to independently transfer from bed to wheelchair with or without aids but without assistance of another person
* Able to understand and communicate in Swedish
* Able to use and access to technical devices for online meetings i.e., computers or tablets with internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Fall Prevention Strategy Survey | Change from baseline in number of strategies used at 18 weeks after the start of the intervention/control period
  The scale includes 14 fall prevention strategies. Participants report whether they currently use or have used the strategies to manage falls risk. If they are using it, they rate strategy effectiveness on a scale of 0-10. If they are not using it, they identify why (e.g., forgot, didn't think it would work, don't know how). The number of strategies used is calculated where a higher number of strategies indicate a better outcome
Fall Prevention Strategy Survey | Number of strategies used at 18 weeks after the start of the intervention/control period
  The scale includes 14 fall prevention strategies. Participants report whether they currently use or have used the strategies to manage falls risk. If they are using it, they rate strategy effectiveness on a scale of 0-10. If they are not using it, they identify why (e.g., forgot, didn't think it would work, don't know how). The number of strategies used is calculated where a higher number of strategies indicate a better outcome

SECONDARY OUTCOMES:
Falls incidence | Weekly from baseline to the 18-week follow-up
  Falls will be monitored via an online short message service (SMS) and interview
Measure of fear of falling | At baseline, and at follow-ups seven and 18 weeks after the start of the intervention/control period
  Questionnaire with one question "Are you afraid of falling?" and six response options: Not at all afraid, Somewhat afraid, Fairly afraid, Very afraid, Don't know, Refused
Falls Efficacy Scale -International | At baseline, and at follow-ups seven and 18 weeks after the start of the intervention/control period
  Questionnaire that consists of 16 questions regarding 'how concerned' the person is when performing daily activities. Each question is answered with a four-graded scale (1-4); not at all concerned, somewhat concerned, fairly concerned and very concerned. A total score is calculated and ranges from 16 to 64
Spinal Cord Injury Fall Concern Scale | At baseline, and at follow-ups seven and 18 weeks after the start of the intervention/control period
  Addresses concern about falling during 16 activities of daily living associated with falling, scored on a 4-point scale (1=not at all concerned to 4=very concerned. The total score is calculated by summing the scores for each activity, with a possible range between 16 and 64
Multiple Sclerosis Impact Scale | At baseline, and at follow-ups seven and 18 weeks after the start of the intervention/control period
  29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of multiple sclerosis on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease
Frenchay Activities Index | At baseline, and at follow-ups seven and 18 weeks after the start of the intervention/control period
  Measures frequency of social and everyday activities. The Frenchay Activities Index consists of 15 items and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Academic Specialist Centre of Neurology, Stockholm
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in a publication, after deidentification.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Immediately following publication and ending two years after publication
Access Criteria: Since data can indirectly be traced back to the study participants, according to the Swedish and EU personal data sharing legislation, access can only be granted upon request. Request for access to the data can be put to our Research Data Office (rdo@ki.se) at Karolinska Institutet, and will be handled according to the relevant legislation. In most cases, this will require a data processing agreement or similar with the recipient of the data.

REFERENCES:
- [Background] Kierkegaard M, Peterson E, Tuvemo Johnson S, Gottberg K, Johansson S, Elf M, Flink M, Ytterberg C. Online self-management fall prevention intervention for people with multiple sclerosis: a feasibility study protocol of a parallel group randomised trial. BMJ Open. 2022 Jul 8;12(7):e061325. doi: 10.1136/bmjopen-2022-061325. PMID 35803627
- [Result] Tuvemo Johnson S, Flink M, Peterson E, Gottberg K, Elf M, Johansson S, Kierkegaard M, Ytterberg C. Self-management of falls in people with multiple sclerosis: A scoping review. Clin Rehabil. 2023 Feb;37(2):162-176. doi: 10.1177/02692155221128723. Epub 2022 Sep 29. PMID 36177511
- [Result] Meijer U, Flink M, Tuvemo Johnson S, Kierkegaard M, Gottberg K, Ytterberg C. Preventing falls in multiple sclerosis: a qualitative study on user requirements for a self-management programme. Disabil Rehabil. 2025 Jan;47(2):398-405. doi: 10.1080/09638288.2024.2348725. Epub 2024 May 7. PMID 38711397
- [Result] Johnson ST, Ytterberg C, Peterson E, Johansson S, Kierkegaard M, Gottberg K, Flink M. Development of Fewer Falls in MS-An Online, Theory-Based, Fall Prevention Self-Management Programme for People With Multiple Sclerosis. Health Expect. 2024 Aug;27(4):e14154. doi: 10.1111/hex.14154. PMID 39032151